CLINICAL TRIAL: NCT01581996
Title: Effect of Lanthanum Carbonate (Fosrenol) on Fecal Phosphorus Excretion and Phosphorus Balance
Brief Title: Fosrenol and Phosphorus Balance - Lanthanum Carbonate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20266-01
Record Dates: First submitted 2012-04-09; First posted 2012-04-20 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Chronic Kidney Failure; End-stage Renal Disease; Disorders Associated With Peritoneal Dialysis
Keywords: Chronic renal failure; End-stage renal disease; Chronic peritoneal dialysis; Serum phosphorus; Hyperphosphatemia; Phosphate binders; Phosphate
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia | interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lanthanum carbonate treatment (Experimental): One Treatment arm. All patients will receive the following doses of lanthanum carbonate(Fosrenol)for 10-12 days each: 0 mg, 500 mg tid, 1000 mg tid and 1500 mg tid.
  Interventions: Drug: lanthanum carbonate

INTERVENTIONS:
Drug: lanthanum carbonate — All patients will receive the following doses of lanthanum carbonate in random order for 10 -12 days each. O mg, 500 mg tid, 1000 mg tid, 1500 mg tid.
  Other Names: Fosrenol

SUMMARY:
Positive phosphorus balance and hyperphosphatemia (increased serum phosphorus levels) are very common complications of people with advanced chronic kidney disease (i.e., stage 5 CKD), including chronic dialysis patients, and are associated with severe morbidity and increased mortality. Despite attempts to control serum phosphorus with dietary phosphorus restriction and the use of medicines that bind phosphorus in the gastrointestinal tract so that the phosphorus cannot be absorbed into the body( also called phosphate binders), chronic dialysis patients frequently remain hyperphosphatemic, particularly at the time when they commence each of their regular dialysis treatments.

Fosrenol (lanthanum carbonate, manufactured by Shire Pharmaceuticals) is a gastrointestinal phosphate binder that appears to have the advantages of being safe, well tolerated and effective at binding phosphate. There are limited data on the magnitude of binding of phosphorus by Fosrenol in the human gastrointestinal tract of patients with chronic kidney disease.

The specific aims for this proposal are as follows:

1. To quantify, under precisely controlled metabolic balance conditions, the increase in fecal excretion of dietary phosphorus that occurs when patients undergoing chronic peritoneal dialysis (CPD) ingest Fosrenol (lanthanum carbonate).
2. To examine a dose response relationship between Fosrenol treatment and fecal phosphorus excretion. The investigators will examine in CPD patients ingesting a constant phosphorus intake, how much additional phosphorus is excreted in the feces at three different dose levels of Fosrenol, 1.5, 3.0, and 4.5 g/day.
3. To examine how increased fecal phosphorus losses and more negative phosphorus balance caused by Fosrenol intake affects serum phosphorus and such hormonal regulators of phosphorus metabolism as serum parathyroid hormone (PTH), fibroblast growth factor-23, 25-hydroxycholecalciferol (25(OH)D3), 1,25-dihydroxycholecalciferol (1,25(OH)2D3) and fetuin-A.
4. To assess whether there is any effect of Fosrenol and increased intestinal phosphate binding on protein-nitrogen balance.

DETAILED DESCRIPTION:
Seven clinically stable patients who have been undergoing CPD for at least six months will be admitted to the General Clinical and Research Center (GCRC) at Harbor-UCLA Medical Center for 46 days. During this time they will be fed, under strict metabolic balance study conditions, a constant energy and protein intake designed to meet their previously ascertained nutritional needs. Their dietary intakes of phosphorus, calcium and magnesium will be maintained constant throughout the 46 days of study at 1100 mg/day, 1000 mg/day and 200 mg/day, respectively. Patients will be treated throughout the study with a constant peritoneal dialysis regimen that consists of either continuous ambulatory peritoneal dialysis with four dialysate exchanges daily or automated peritoneal dialysis in which they will each receive about four dialysate exchanges per night; and possibly day-time dialysate exchanges. The number and volume of dialysate exchanges and the dialysate glucose concentration may vary among patients according to their metabolic and clinical needs, but will be constant for each patient. Patients will adhere to standard metabolic balance protocols as the investigators have conducted during our many previous metabolic balance studies. These protocols will include participating in prescribed daily exercise regimens that are designed to maintain the patients' physical activity at their prestudy, outpatient levels.

All patients will first undergo a 10 day Baseline period for metabolic equilibration during which time they will not receive any phosphate binder. They will then receive three periods of Fosrenol treatment with three different dose levels for 12 days each. During each of three periods, the patients will receive, in random order, one or two Fosrenol tablets that will provide 500, 1000, or 1500 mg with each of the three meals that they will be fed each day. Thus these CPD patients will receive in random order 1500, 3000 and 4500 mg/day of Fosrenol each prescribed for one 12 day period.

Outcome Measurements. All urine, collected in 24 hour urine specimens, and all feces excreted, collected over four day periods, will be obtained continuously. Every 4 days a duplicate 24 hour diet will be prepared for chemical analyses. The above specimens will be analyzed for phosphorus, calcium and nitrogen by spectrographic, atomic absorption spectroscopic and Kjeldahl analyses, respectively. Serum phosphorus, calcium, parathyroid hormone (PTH), fibroblast growth factor-23, 25-hydroxycholecalciferol (25(OH)D3), 1,25-dihydroxycholecalciferol (1,25(OH)2D3), fetuin-A, urea and creatinine will be measured in the fasting state at the beginning of the 40 day balance period and every 5 days. Anthropometry and other standard measurements that are routinely conducted during metabolic balance procedures will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Chronic peritoneal dialysis treatment(CPD) for at least the previous six months, Clinically stable,
* Ages 30 to 65 years old,
* Both genders,
* Any racial or ethnic background,
* Evidence that the subject is capable of giving informed consent and of adhering to the study protocol.

Exclusion Criteria:

* No inflammatory or catabolic illnesses.
* No hospitalizations within the previous three months except for vascular access revision,
* No severe heart, liver or lung failure,
* No cancer, other than basal cell carcinoma, systemic infections, vasculitis or other rheumatological diseases.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Fecal Phosphorus and Body Phosphorus Balance | Two years
  Dose response relationship between lanthanum carbonate(Fosrenol) intake and fecal phosphorus excretion and body phosphorus balance. Specifically, the phosphorus content of feces, urine, expended dialysate, diet and any vomitus or rejected food will be measured.

SECONDARY OUTCOMES:
Fecal Calcium and Nitrogen and Body Calcium and Nitrogen Balance | Two years
  Fecal calcium and nitrogen and calcium and nitrogen balance in chronic peritoneal dialysis patients eating lanthanum carbonate (Fosrenol) intake. Effect of ingestion of Fosrenol on serum phosphorus and hormonal regulators of phosphorus metabolism as serum, parathyroid hormone (PTH), fibroblast growth factor-23, 25-hydroxycholecalciferol (25(OH)D3), 1,25-dihydroxycholecalciferol (1,25(OH)2D3) and fetuin-A.
Protein-nitrogen balance | Two years
  Lanthanum carbonate (Fosrenol) and increased intestinal phosphate binding on protein-nitrogen balance.
Gastrointestinal symptoms | Two years
  Gastrointestinal symptoms, particularly for anorexia, nausea vomiting, abdominal pain, distention, flatulence, constipation, diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Joel D. Kopple, M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

REFERENCES:
- [Derived] Kopple JD, Bross R, Ekramzadeh M, Markovic D, Lyzlov A, Lodebo BT, Mehrotra R, Shah AP. Lanthanum carbonate lowers serum phosphorus without altering body phosphorus burden in maintenance peritoneal dialysis patients: a randomized crossover trial. Am J Clin Nutr. 2025 Dec;122(6):1858-1868. doi: 10.1016/j.ajcnut.2025.08.015. Epub 2025 Oct 1. PMID 41033875